CLINICAL TRIAL: NCT02768974
Title: An Open Label, Proof of Concept Study to Assess the Safety, PK and Explore Efficacy of OPRX-106 in Patients With Active Mild to Moderate Ulcerative Colitis
Brief Title: Open Label Study to Assess Safety, PK and Explore Efficacy of OPRX-106 in Patients With Active Mild to Moderate Ulcerative Colitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Protalix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PB-106-003
Record Dates: First submitted 2016-03-27; First posted 2016-05-11 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-05

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OPRX-106 2 mg (Experimental): Open label, 1:1 randomization ration (up to 10 subjects)
  Interventions: Drug: OPRX-106
- OPRX-106 8 mg (Experimental): Open label, 1:1 randomization ration (up to 10 subjects)
  Interventions: Drug: OPRX-106

INTERVENTIONS:
Drug: OPRX-106 — Oral delivery, once daily.

SUMMARY:
This is a proof of concept, randomized, open label, 2-arm study of OPRX-106 in subjects with active mild to moderate ulcerative colitis. Eligible subjects will be enrolled and randomized to receive 2 mg or 8 mg of OPRX-106 administered orally, once daily for 8 weeks.

ELIGIBILITY:
Main Inclusion Criteria:

1. Have had a diagnosis of ulcerative colitis for a minimum of 3 months
2. Have active mild to moderate ulcerative colitis, as defined by a full Mayo score at screening
3. Have adequate cardiac, renal and hepatic functions as determined by the investigator and demonstrated by screening clinical and laboratory evaluations, and physical examination results
4. High level of calprotectin (>100 mg/kg of stool)

Main Exclusion Criteria:

1. Have a history of colonic or rectal surgery other than hemorrhoidal surgery or appendectomy
2. .Positive for active/ latent mycobacterium tuberculosis (TB) infection
3. .Have a history of infection requiring administration of any IV antibiotic, antiviral or antifungal medication or any oral anti-infective agent
4. Severe ulcerative colitis
5. Ulcerative proctitis, defined as disease limited to less than 15 cm from the anal verge
6. Use >4.8 g 5-ASA or equivalent
7. Use of corticosteroid or 5-ASA enemas, foams, or suppositories
8. Use of anti-inflammatory medications or natural remedies
9. Use oral or parenteral antibiotics
10. Use of chronic non-steroidal anti-inflammatory (NSAID) therapy
11. Use of immune suppressive agents including anti-TNF agents, Azathioprine, 6MP, Methotrexate
12. Use of steroids
13. Have a diagnosis of: Crohn's disease; Indeterminate colitis; Microscopic colitis; Ischemic or infectious colitis; Clostridium difficile colitis, Parasitic disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Adverse events following daily administration of OPRX 106 | 70 days
  Adverse events from subject reporting or other assessments

OTHER OUTCOMES:
OPRX-106 individual plasma levels following single and multiple dose administrations | 56 days
Clinical response or clinical remission from baseline to end of OPRX 106 treatment | Baseline to day 56
  Based on Mayo score
Histopathological improvement (Geboes scale) from baseline to end of OPRX treatment | Baseline to day 56
Improvement from baseline to end of OPRX 106 treatment in hs-CRP levels | Baseline to day 56
Improvement from baseline to end of OPRX 106 treatment in fecal calprotectin levels | Baseline to day 56

CONTACTS AND LOCATIONS:
Overall Officials: Einat Dekel, DVM, Study Director — Sr. Director Clinical Development
Locations (7):
- Israel (7):
  - Soroka University Hospital, Beersheba
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Center, Jerusalem
  - Shaare-Zedek Medical Center, Jerusalem
  - Galilee Medical Center, Nahariya
  - Assaf-Harofeh Medical Center, Rishon LeZiyyon
  - Tel-Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: Undecided